CLINICAL TRIAL: NCT05611996
Title: PEERS Plus - mHealth Enhanced Peer Support to Reduce Depression Among Low-income and Ethnic Minority Older Adults
Brief Title: PEERS Plus mHealth Enhanced Peer Support
Acronym: Peers plus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jin hui Joo, MD, MA, Assistant Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022P001984
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Results first posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Depression in Old Age

STUDY DESIGN:
Intervention Model Description: A cohort of 20 older adults will be assigned to the Peer plus program for 8 weeks, without a comparison group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peer support (Other): Peer mentors who have experienced depression provide social support through video chats and texts for 8 weeks.
  Interventions: Behavioral: Peers plus

INTERVENTIONS:
Behavioral: Peers plus — Peer support intervention in which peer mentors who have experiential knowledge of depression deliver social support through video chats and texts to older adults with depression.

SUMMARY:
The goal of this intervention study is to design and learn whether peer support that is delivered through video chats and texts can decrease depression among older adults. Participants will be assigned to a peer support program where they will receive 8 video chats with a peer mentor who provide social support and supportive texts over 8 weeks.

DETAILED DESCRIPTION:
PEERS plus is a psychosocial intervention being developed to reduce depression among older adults. In this intervention peer mentors who are also 50 years of age and older and who have experiential knowledge of depression provide depression care. Older adults with depression will be recruited and assigned to the peer support program. This will consist of 8 weekly peer mentor - older adult video chats that provide emotional support and sharing of self-care skills for depression. Supportive texts will be sent on a weekly basis to older adults by peer mentors. These texts will provide encouragement, affirmations and information about mental health resources. Peer mentors are trained and supervised by a mental health professional during the 8 week period. We will assess at baseline, post study and 3 months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. 50 years and older
2. PHQ-9 score > 5,
3. on the same antidepressant dose for at least 3 months
4. if receiving psychotherapy, frequency is at most once a month
5. able to communicate in English
6. able to give informed consent.

Exclusion Criteria:

1. meet diagnostic criteria for mania or hypomania
2. active suicidal ideation
3. meet diagnostic criteria for psychotic syndrome
4. meet diagnostic criteria for substance abuse or dependence
5. cognitive impairment, with a score on the Short Blessed Test > 9.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Peer Support: Older adults who are experiencing depression receive peer support. Peer support consists of emotional and self care support delivered by a peer mentor. Peer mentors are the interventionists and do not receive the intervention. We did not collect any data about peer mentors in the study.
Period: Overall Study
Arm/Group | Peer Support
Started | 34
Completed | 24
Not Completed | 10
Not completed — Ineligible | 1
Not completed — Withdrawal by Subject | 9

BASELINE CHARACTERISTICS:
Population: Peer mentors who have experienced depression provide social support through video chats and texts for 8 weeks.
  Peers plus: Peer support intervention in which peer mentors who have experiential knowledge of depression deliver social support through video chats and texts to older adults with depression.
  Baseline data were not collected from peer mentors participants and peer mentors were not assessed for adverse events.
Arm/Group | Peer Support
Number analyzed (Participants) | 34
Age, Continuous [Mean (Full Range); unit: years] — Population: 34 participants started the intervention, 28 finished the intervention and 6 dropped during the intervention.
  years | 66.62 [50 to 84]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 34 participants started the intervention, 28 finished the intervention and 6 dropped during the intervention.
  Participants
    Female | 31
    Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 34 participants started the intervention, 28 finished the intervention and 6 dropped during the intervention.
  Participants
    Hispanic or Latino | 1
    Not Hispanic or Latino | 33
    Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 34 participants started the intervention, 28 finished the intervention and 6 dropped during the intervention.
  Participants
    Asian | 2
    Black | 9
    White | 21
    Multiracial | 2
Region of Enrollment [Count of Participants; unit: Participants] — Population: 34 participants started the intervention, 28 finished the intervention and 6 dropped during the intervention.
  Participants
    United States | 34
Patient Health Questionnaire-9 [Mean (Standard Deviation); unit: units on a scale] — Depression will be assessed with the Patient Health Questionnaire (PHQ-9). The PHQ-9 score is summed from 9 items in the questionnaire, and scores range from 0 to 27. A higher score indicates a worse outcome in depression. A score of 5 indicates mild depressive symptoms, 10 - 14 indicates moderate depression, 15-19 indicates moderately severe depression, and 20-27 indicates severe depression. Population: 34 participants started the intervention, 28 finished the intervention and 6 dropped during the intervention.
  units on a scale | 11.32 (5.36)

OUTCOME MEASURES:

1. Primary Outcome: Intervention Feasibility
Description: Proportion of the participants who complete 80% of their weekly meetings with the peer coach.
Time Frame: 18 months
Population: Peer mentors who have experienced depression provide social support through video chats and texts for 8 weeks.
  Peers plus: Peer support intervention in which peer mentors who have experiential knowledge of depression deliver social support through video chats and texts to older adults with depression.
Measure: Count of Participants; unit: Participants
Arm/Group | Peer Support
Number analyzed (Participants) | 34
Participants | 28

2. Other Pre Specified Outcome: Patient Health Questionnaire-9
Description: Depression will be assessed with the Patient Health Questionnaire (PHQ-9). The PHQ-9 score is summed from 9 items in the questionnaire, and scores range from 0 to 27. A higher score indicates a worse outcome in depression. A score of 5 indicates mild depressive symptoms, 10 - 14 indicates moderate depression, 15-19 indicates moderately severe depression, and 20-27 indicates severe depression.
Time Frame: We assessed PHQ-9 scores as changes across three timepoints: baseline, post study and 3 month follow up. We ran a mixed-effects longitudinal model to examine how PHQ-9 scores changed over 5 months (8 week intervention and 3 month follow up).
Population: Sample sizes varied across the three timepoints due to participant attrition. Some individuals chose not to proceed with the intervention after completing the baseline assessment, while others were lost to follow-up by the post-intervention or 3-month follow-up assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peer Support
Number analyzed (Participants) | 34
score on a scale
  Baseline | 11.32 (5.36)
  Post Study: number analyzed (Participants) | 28
  Post Study | 9.71 (5.59)
  3 Month Follow Up: number analyzed (Participants) | 24
  3 Month Follow Up | 8.29 (4.84)
Statistical Analysis 1: Comparison: Peer Support; Null hypothesis: there is no difference in the mean Patient Health Questionnaire-9 (PHQ-9) scores from baseline to post-intervention for all study participants; Test type: Superiority; p = 0.025, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Mean Difference (Net) = -1.783, 95% CI 2-sided [-3.336 to -0.230], Standard Error of Mean 0.772 — Score difference = Post-intervention - Baseline
Statistical Analysis 2: Comparison: Peer Support; Null hypothesis: there is no difference in the mean Patient Health Questionnaire-9 (PHQ-9) scores from baseline to 3-month for all study participants; Test type: Superiority; p = 0.005, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Mean Difference (Net) = -2.420, 95% CI 2-sided [-4.057 to -0.784], Standard Error of Mean 0.814 — Score difference = 3-month - Baseline
Statistical Analysis 3: Comparison: Peer Support; Null hypothesis: There is no difference in the mean Patient Health Questionnaire-9 (PHQ-9) scores over time for all study participants; Test type: Superiority; p = 0.0040, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Mean Difference (Net) = -0.5468, 95% CI 2-sided [-0.9039 to -0.1897], Standard Error of Mean 0.1744 — The mean difference of the PHQ-9 score by each unit increase of the time(each week increase)

ADVERSE EVENTS:
Time Frame: Adverse event data is collected through study completion, an average of 18 months.
Description: Baseline data were not collected from peer mentors and peer mentors were not assessed for adverse events.
Arm/Group | Peer Support
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-08-07): https://cdn.clinicaltrials.gov/large-docs/96/NCT05611996/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT05611996/SAP_001.pdf